CLINICAL TRIAL: NCT03913715
Title: Ostomy Rural Telehealth Self-management Training for Cancer Survivors
Brief Title: Ostomy Rural Telehealth Training Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 832343; R01CA204193 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-04-12 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ostomy; Quality of Life; Telehealth
Keywords: Ileostomy, Urostomy, Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ostomy Self-Management Training (Active Comparator): Ostomy Self-management Training group in which subject will learn using pouches and equipment, skincare, ostomy complications, nutritional needs, Impact on feelings, clothing changes, social relationships, being prepared for emergencies, Intimacy and sexuality, communication skills, tips for traveling and physical activity recommendations
  Interventions: Other: Ostomy Self-Management Training
- Usual care (Placebo Comparator): Usual care in peri-operative and long-term settings is not standardized for ostomy patients. Usual care does not provide any formal, reproducible training for patients or their caregivers. It typically consists of an Ostomy Care Nurse who works with patients and caregivers concerning technical issues (fitting, emptying, supplies, surrounding skin care, etc.) while the new ostomate is still an inpatient.
  Interventions: Other: Ostomy Self-Management Training

INTERVENTIONS:
Other: Ostomy Self-Management Training — Ostomy Self management Training group in which subject will learn using pouches and equipment, skincare, ostomy complications, nutritional needs, Impact on feelings, clothing changes, social relationships, being prepared for emergencies, Intimacy and sexuality, communication skills, tips for traveling and physical activity recommendations

SUMMARY:
Over one million individuals in the U.S. have ostomies. The American Cancer Society estimates 43,030 rectal cancer cases and 81,190 bladder cancer cases will be diagnosed in 2018.Of these, at least 30,000 will receive ostomies, and an additional unknown number due to gynecologic, other gastrointestinal, or other gastro-urinary tumors. The health-related quality of life impact is tremendous and greater than with many other cancer treatments. An ostomy is often a prolonged or lifelong disabling problem for cancer survivors. The adaptation period is quite variable. In our R01 study, 18% of participants took at least one year to be comfortable, or never felt comfortable, in managing their ostomy care. Importantly, many patients cannot attend in-person self-management programs or patient groups for a myriad of reasons, including distance to travel, lack of access to transportation, monetary outlays, competing demands (such as work), or comorbidities making travel difficult. In addition, a national shortage of OCNs means patients with an ostomy, whether newly placed or a long-term issue, receive little help. It is imperative to study interventions for rural survivors aimed to limit family financial burdens, improve ostomy outcomes, and improve survivors' well-being.

DETAILED DESCRIPTION:
An ostomy adversely affects health-related quality of life in a diverse population of cancer survivors. For cancer, ostomies are most commonly placed for rectal cancers, followed by urinary bladder cancer. Ostomies may be needed for other cancers related to bulky or metastatic disease, or in emergencies. In addition, ostomies may be placed on a temporary or a permanent basis. Temporary ostomies may be created in emergencies, such as perforation or obstruction due to tumor, or in planned procedures, as with a low rectal resection for cancer where an ostomy is placed to "protect" a new anastomosis while it heals. Temporary ostomies may become permanent as a result of underlying comorbidities, need for other treatments related to cancer, or poor outcome of anastomosis (leak or stricture). Peri-operative needs are the same regardless of ostomy permanence; survivors should receive clear, systematic, evidence-based ostomy self-management instruction and support.

To cope with the challenges of their diseases, cancer survivors with ostomies should have confirmed levels of self-management skills, as well as strong commitments to self-management. Cognitive restructuring, problem-solving, and self-efficacy/locus of control are essential tools for effective self-management. As in most chronic conditions, this tends to be long-term, complex, and multidimensional. Trial-and-error ostomy self-care, nurse counseling, and community referral have been the primary modes of self-management education and support in the peri-operative period. Clearly, ostomates face many obstacles in coping with their condition, not least of which is medical care that often does not meet their needs for effective information, clinical management, psychological support, and patient activation These obstacles are likely compounded for ostomates living in rural areas. Approximately 14-19% of the US population resides in rural areas. Rural cancer survivors face significant barriers to ongoing care including lack of access to specialists and cancer-specific specialized support, longer travel distances to access follow-up care, and transportation challenges due to financial barriers or lack of a vehicle. Individuals in rural areas travel a median of 51-59 minutes to reach specialized oncology care. Additionally, some studies suggest that rural cancer patients have worse quality of life and mental health than their urban counterparts, and up to a quarter of rural cancer patients have unmet cancer information needs. Telehealth delivery of an ostomy self-management program offers an opportunity to reduce these access disparities among rural ostomates.

Ostomates and their families must engage in ostomy self-management, make behavior changes, and adjust to the consequences of their condition, becoming the principal caretakers and navigators. Preparation of the survivor and unpaid designated caregiver/support person (usually family members) is requisite to assure optimal functioning and HRQOL, as well as to prevent or ameliorate ostomy-related complications and associated health care utilization. Multiple communication issues make it difficult for ostomy survivors to access resources for improving their self-management, and undermine opportunities to improve and sustain HRQOL. These resources include lack of consistent follow-up, travel issues, lack of surgeon focus on ostomy-related problems, and lack of ostomy nurse clinic resources.

Ostomies are associated with multiple HRQOL difficulties. Ongoing problems include pouching care, travel out of the home (especially relevant for rural populations), social interactions, intimacy, and acceptance of/satisfaction with appearance. Studies document persistent challenges including sexuality psychological problems and interference with work, recreation, and sporting activities. However, improved self-efficacy eases the psychological and social burden of ostomies. No reports have been published on the results of a systematic ostomy self-management program to ensure optimal post-operative care, including adaptation, self-management, and ostomy comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer or pre-cancer (e.g. carcinoma in situ or severe dysplasia) survivors over 18 years of age having undergone a procedure that needed an intestinal stoma (fecal or urinary). Survivors with temporary ostomies will be included.
2. Residence within a zip code that is designated as non-metropolitan or non-urban.
3. All participants must have a full understanding of the protocol and be able to sign an informed consent form.
4. Participants must be able to complete the study questionnaires and sessions in English.
5. Having an identified caregiver/support person is NOT a requirement for eligibility but will be strongly encouraged if possible.
6. All participants will attend their first training session at least six weeks after their operation.
7. There is no maximum time since surgery.
8. Eligible patients with temporary ostomies must NOT undergo ostomy reversal:

   i. While they are participating in the training sessions (intervention arm). ii. During the corresponding time of the training sessions (usual care arm)
9. Subjects must be willing to complete the surveys described in the protocol.

Exclusion Criteria:

* N/A

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient Activation - PAM | 0 months
  Patient Activation Measure. It uses a uni-dimensional, probabilistic Guttman-like scale that reflects a developmental model of activation that involves four stages: (1) believing the patient role is important, (2) having the confidence and knowledge necessary to take action, (3) actually taking action to maintain and improve one's health, and (4) staying the course even under stress. The measure can be used at the individual patient level to tailor interventions and assess changes. Those with higher activation scores report significantly better health, and significantly lower rates of doctor office visits, emergency room visits, and hospital nights. High internal consistency and construct validity have been reported.
Patient Activation- PAM | 2 months
  Patient Activation Measure. It uses a uni-dimensional, probabilistic Guttman-like scale that reflects a developmental model of activation that involves four stages: (1) believing the patient role is important, (2) having the confidence and knowledge necessary to take action, (3) actually taking action to maintain and improve one's health, and (4) staying the course even under stress. The measure can be used at the individual patient level to tailor interventions and assess changes. Those with higher activation scores report significantly better health, and significantly lower rates of doctor office visits, emergency room visits, and hospital nights. High internal consistency and construct validity have been reported.
Patient Activation - PAM | 3 months
  Patient Activation Measure. It uses a uni-dimensional, probabilistic Guttman-like scale that reflects a developmental model of activation that involves four stages: (1) believing the patient role is important, (2) having the confidence and knowledge necessary to take action, (3) actually taking action to maintain and improve one's health, and (4) staying the course even under stress. The measure can be used at the individual patient level to tailor interventions and assess changes. Those with higher activation scores report significantly better health, and significantly lower rates of doctor office visits, emergency room visits, and hospital nights. High internal consistency and construct validity have been reported.
Patient Activation- PAM | 6 months
  Patient Activation Measure.It uses a uni-dimensional, probabilistic Guttman-like scale that reflects a developmental model of activation that involves four stages: (1) believing the patient role is important, (2) having the confidence and knowledge necessary to take action, (3) actually taking action to maintain and improve one's health, and (4) staying the course even under stress. The measure can be used at the individual patient level to tailor interventions and assess changes. Those with higher activation scores report significantly better health, and significantly lower rates of doctor office visits, emergency room visits, and hospital nights. High internal consistency and construct validity have been reported.
Patient Activation- PAM | 12months
  Patient Activation Measure.It uses a uni-dimensional, probabilistic Guttman-like scale that reflects a developmental model of activation that involves four stages: (1) believing the patient role is important, (2) having the confidence and knowledge necessary to take action, (3) actually taking action to maintain and improve one's health, and (4) staying the course even under stress. The measure can be used at the individual patient level to tailor interventions and assess changes. Those with higher activation scores report significantly better health, and significantly lower rates of doctor office visits, emergency room visits, and hospital nights. High internal consistency and construct validity have been reported.

SECONDARY OUTCOMES:
Self-efficacy | 0 months
  Self-Efficacy to Perform Ostomy Self-Management Behaviors.Modified from Lorig and colleagues' Self-Efficacy to Perform Self-management Behaviors Scale, an outcome measure for Chronic Disease Management Interventions, this scale represents 8 domains (with reported Cronbach's alpha for original scales,physical activity , information seeking, support, communication with HC providers, ostomy management, social and recreational, symptom management and depression.
Self-efficacy | 2 months
  Self-Efficacy to Perform Ostomy Self-Management Behaviors.Modified from Lorig and colleagues' Self-Efficacy to Perform Self-management Behaviors Scale, an outcome measure for Chronic Disease Management Interventions, this scale represents 8 domains (with reported Cronbach's alpha for original scales,physical activity , information seeking, support, communication with HC providers, ostomy management, social and recreational, symptom management and depression.
Self-efficacy | 6 months
  Self-Efficacy to Perform Ostomy Self-Management Behaviors.Modified from Lorig and colleagues' Self-Efficacy to Perform Self-management Behaviors Scale, an outcome measure for Chronic Disease Management Interventions, this scale represents 8 domains (with reported Cronbach's alpha for original scales,physical activity , information seeking, support, communication with HC providers, ostomy management, social and recreational, symptom management and depression.
Self-efficacy | 12 months
  Self-Efficacy to Perform Ostomy Self-Management Behaviors.Modified from Lorig and colleagues' Self-Efficacy to Perform Self-management Behaviors Scale, an outcome measure for Chronic Disease Management Interventions, this scale represents 8 domains (with reported Cronbach's alpha for original scales,physical activity , information seeking, support, communication with HC providers, ostomy management, social and recreational, symptom management and depression.
Health-related quality of life | 0 months
  COH-QOL-CRC Scale.The City of Hope QOL-Ostomy questionnaire was designed for all adult ostomates, and has a 4-dimensional HRQOL (physical, psychological, social and spiritual well-being) framework gathering demographic, personal (e.g. diet, work, and activity) and clinical data. It has an open-ended question of the greatest challenge of ostomy survivors. A multi-item scale section assesses overall Health-related quality of life and the four Health-related quality of life dimensions on a 0 to 10 scale. The full survey will be used at baseline; for post intervention and follow-up, only the 43 scaled items (those items sensitive to change over time) will be used. Reported Cronbach's alphas are .94 total scale and .80-.90 subscales.
Health-related quality of life | 2 months
  COH-QOL-CRC Scale.The City of Hope QOL-Ostomy questionnaire was designed for all adult ostomates, and has a 4-dimensional HRQOL (physical, psychological, social and spiritual well-being) framework gathering demographic, personal (e.g. diet, work, and activity) and clinical data. It has an open-ended question of the greatest challenge of ostomy survivors. A multi-item scale section assesses overall Health-related quality of life and the four Health-related quality of life dimensions on a 0 to 10 scale. The full survey will be used at baseline; for post intervention and follow-up, only the 43 scaled items (those items sensitive to change over time) will be used. Reported Cronbach's alphas are .94 total scale and .80-.90 subscales.
Health-related quality of life | 3 months
  COH-QOL-CRC Scale.The City of Hope QOL-Ostomy questionnaire was designed for all adult ostomates, and has a 4-dimensional HRQOL (physical, psychological, social and spiritual well-being) framework gathering demographic, personal (e.g. diet, work, and activity) and clinical data. It has an open-ended question of the greatest challenge of ostomy survivors. A multi-item scale section assesses overall Health-related quality of life and the four Health-related quality of life dimensions on a 0 to 10 scale. The full survey will be used at baseline; for post intervention and follow-up, only the 43 scaled items (those items sensitive to change over time) will be used. Reported Cronbach's alphas are .94 total scale and .80-.90 subscales.
Health-related quality of life | 6 months
  COH-QOL-CRC Scale.The City of Hope QOL-Ostomy questionnaire was designed for all adult ostomates, and has a 4-dimensional HRQOL (physical, psychological, social and spiritual well-being) framework gathering demographic, personal (e.g. diet, work, and activity) and clinical data. It has an open-ended question of the greatest challenge of ostomy survivors. A multi-item scale section assesses overall Health-related quality of life and the four Health-related quality of life dimensions on a 0 to 10 scale. The full survey will be used at baseline; for post intervention and follow-up, only the 43 scaled items (those items sensitive to change over time) will be used. Reported Cronbach's alphas are .94 total scale and .80-.90 subscales.
Health-related quality of life | 12 months
  COH-QOL-CRC Scale.The City of Hope QOL-Ostomy questionnaire was designed for all adult ostomates, and has a 4-dimensional HRQOL (physical, psychological, social and spiritual well-being) framework gathering demographic, personal (e.g. diet, work, and activity) and clinical data. It has an open-ended question of the greatest challenge of ostomy survivors. A multi-item scale section assesses overall Health-related quality of life and the four Health-related quality of life dimensions on a 0 to 10 scale. The full survey will be used at baseline; for post intervention and follow-up, only the 43 scaled items (those items sensitive to change over time) will be used. Reported Cronbach's alphas are .94 total scale and .80-.90 subscales.
Ostomy knowledge | 0 months
  Ostomy Knowledge Questionnaire.This brief survey, derived at City of Hope, was modified for the pilot study and further adapted by the study team to ensure major topics were included.
Ostomy knowledge | 2 months
  Ostomy Knowledge Questionnaire.This brief survey, derived at City of Hope, was modified for the pilot study and further adapted by the study team to ensure major topics were included.
Ostomy knowledge | 6 months
  Ostomy Knowledge Questionnaire.This brief survey, derived at City of Hope, was modified for the pilot study and further adapted by the study team to ensure major topics were included.
Ostomy knowledge | 12 months
  Ostomy Knowledge Questionnaire.This brief survey, derived at City of Hope, was modified for the pilot study and further adapted by the study team to ensure major topics were included.
Healthcare utilization long form | 0 months
  Based on the model developed by Given, et al., for long-term care, this survey will gather participant self-reports of ostomy-related medical care use, productivity losses, and associated out-of-pocket expenses and time spent for ostomy care in general, and the OSMT intervention, caregivers, and paid housekeeping
Healthcare utilization long form | 6 months
  Based on the model developed by Given, et al., for long-term care, this survey will gather participant self-reports of ostomy-related medical care use, productivity losses, and associated out-of-pocket expenses and time spent for ostomy care in general, and the OSMT intervention, caregivers, and paid housekeeping
Healthcare utilization long form | 12 months
  Based on the model developed by Given, et al., for long-term care, this survey will gather participant self-reports of ostomy-related medical care use, productivity losses, and associated out-of-pocket expenses and time spent for ostomy care in general, and the OSMT intervention, caregivers, and paid housekeeping
Healthcare utilization short form | 2 months
  Based on the model developed by Given, et al., for long-term care, this survey will gather participant self-reports of ostomy-related medical care use, productivity losses, and associated out-of-pocket expenses and time spent for ostomy care in general, and the OSMT intervention, caregivers, and paid housekeeping
Healthcare utilization short form | 3 months
  Based on the model developed by Given, et al., for long-term care, this survey will gather participant self-reports of ostomy-related medical care use, productivity losses, and associated out-of-pocket expenses and time spent for ostomy care in general, and the OSMT intervention, caregivers, and paid housekeeping

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale | 0 months
  Hospital Anxiety and Depression Scale. It is a self-assessment instrument for detecting anxiety and depression in medical outpatients, which has been demonstrated sensitive in community and inpatient cancer studies, with subscales of < 7 not present, 8-10 doubtful, >11 definite. Reported Cronbach's alpha.
Hospital Anxiety and Depression Scale | 2 months
  Hospital Anxiety and Depression Scale. It is a self-assessment instrument for detecting anxiety and depression in medical outpatients, which has been demonstrated sensitive in community and inpatient cancer studies, with subscales of < 7 not present, 8-10 doubtful, >11 definite. Reported Cronbach's alpha.
Hospital Anxiety and Depression Scale | 6 months
  Hospital Anxiety and Depression Scale. It is a self-assessment instrument for detecting anxiety and depression in medical outpatients, which has been demonstrated sensitive in community and inpatient cancer studies, with subscales of < 7 not present, 8-10 doubtful, >11 definite. Reported Cronbach's alpha.
Hospital Anxiety and Depression Scale | 12 months
  Hospital Anxiety and Depression Scale. It is a self-assessment instrument for detecting anxiety and depression in medical outpatients, which has been demonstrated sensitive in community and inpatient cancer studies, with subscales of < 7 not present, 8-10 doubtful, >11 definite. Reported Cronbach's alpha.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krouse, MD, Principal Investigator — University of Pennsylvania
Locations (10):
- United States (10):
  - University of Arkansas For Medical Sciences, Little Rock, Arkansas
  - City Of Hope, Duarte, California
  - Loma Linda University Health, Loma Linda, California
  - University of New Mexico, Albuquerque, New Mexico
  - University of North Carolina, Chapel Hill, North Carolina
  - Sanford Research Center, Fargo, North Dakota
  - Geisinger, Danville, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Medicine, Philadelphia, Pennsylvania
  - University of South Carolina Greenville (Prisma Health), Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code